CLINICAL TRIAL: NCT05741060
Title: Arterial Stiffness, Cognition and Equol
Brief Title: Effect of Equol Supplementation on Arterial Stiffness and Cognition in Healthy Volunteers
Acronym: ACE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akira Sekikawa (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Akira Sekikawa, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY22010165; R01AG074971 (NIH)
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Arterial Stiffness; White Matter Lesions; Cognitive Decline
Keywords: s-equol; white matter lesion volume; vascular contributions to cognitive impairment and dementia; arterial stiffness; Alzheimer's disease and related dementias; estrogen receptor-beta agonist
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease | interventions — Equol

STUDY DESIGN:
Intervention Model Description: The ACE Trial is an early stage multi-center randomized, parallel, double-blind placebo-controlled trial of 10 mg/day of equol for 24 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Equol Arm (Experimental): S-equol - 10 mg per day tablet for 24 months.
  Interventions: Drug: S-equol
- Placebo Arm (Placebo Comparator): 10 mg per day for 24 months of tablets that will be of the same size/shape/color as the experimental tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-equol — Experimental drug
  Other Names: Equelle
  Arms: Equol Arm
Drug: Placebo — Placebo - 10 mg per day for 24 months of tablets that will be the same size/shape/color as the s-equol tablets.
  Arms: Placebo Arm

SUMMARY:
The ACE Trial, funded by the National Institute on Ageing/National Institutes of Health (NIH), is a multicenter clinical trial. The ACE Trial will determine if taking the dietary supplement Equol could slow the progression of stiffening of the arteries, small blood vessel disease in the brain and memory decline. Equol is a soy-based supplement that has plant estrogen-like compounds in it.

Equol is a metabolite of soy isoflavone. Our studies in Japan and other studies suggest that Equol may slow mechanisms related to memory decline. No previous studies in the United States have tested the effect of Equol on these mechanisms or memory decline. Supplementation of Equol in the ACE Trial is approved by the Food and Drug Administration (FDA).

Researchers at the University of Pittsburgh, Pittsburgh, Pennsylvania, Wake Forest University, Winston-Salem, North Carolina, and Emory University, Atlanta, Georgia, are recruiting participants.

The ACE Trial will ask participants to complete 7 clinic visits over a two-year period. The participants are asked to take Equol tablets daily for 24 months. Clinic procedures include Pulse Wave Velocity (to measure arterial stiffness), Magnetic Resonance Imaging (MRI) of the brain and tests of awareness and thinking.

DETAILED DESCRIPTION:
The ACE trial is an early-stage multi-center randomized controlled trial (RCT) designed to test the effect of a 24-month intervention of 10 mg/day equol supplementation on arterial stiffness, white matter lesions (WMLs) in the brain and cognitive decline among 400 individuals aged 65 and 85 without dementia. Recent studies in Japan reported that a diet high in soy and soy isoflavones is inversely associated with incident cognitive impairment and dementia. The Women's Isoflavone Soy Health (WISH) in the US, an RCT of soy isoflavones, however, showed no significant effect on cognition. We posit that the discrepant result is due to the difference in equol-producing capability. Equol, a metabolite of soy isoflavone daidzein transformed by the gut microbiome, is the most bioactive among all soy isoflavones and their metabolites. 50-70% of Japanese convert daidzein to equol in contrast to 20-30% of Americans. Arterial stiffness, a significant predictor of cognitive decline, is significantly improved in a short-duration RCT of 10 mg/day equol supplementation in middle-aged subjects. WMLs are a risk factor for age-related cognitive decline and dementia. We reported a longitudinal association of equol-producing status with WML% (WML volume normalized to total brain volume) in cognitively normal elderly in Japan. The subgroup analysis of WISH showed that equol producers had better cognition than the control group, suggesting that equol may slow cognitive decline. No previous study has tested the effect of equol supplementation on arterial stiffness, WMLs or cognitive decline in older adults.

ELIGIBILITY:
Inclusion Criteria:

Men and women age between 65 and 85 at entry of European Americans or African Americans

Inclusion criteria via screening visit:

* Individuals who are able to provide informed consent
* Individuals who are willing to be randomized to the intervention or placebo group

Exclusion Criteria:

Exclusion criteria via initial screening by phone

* Individuals who are regularly taking isoflavone supplements or eat soy product ≥ 2 times a week (by specific questionnaire)
* Individuals who do not agree to maintain isoflavone supplements or soy product intake described above during the study period.
* Individuals who have allergy or intolerance to soy isoflavones.
* Individuals whose score for the Telephone Interview for Cognitive Status is 22 and below.
* Individuals with stroke, neurological disorders, bipolar disease whether or not under medical treatment, cancer treatment in the past 6 months, head trauma or other condition which is not appropriate for the study (e.g., contraindication to magnetic resonance imaging (MRI)).
* Individuals with untreated depression
* Individuals with atrial fibrillation
* Individuals with heart failure
* Individuals with heart attack or coronary intervention in the past 6 months
* Individuals with carotid endarterectomy or peripheral artery disease
* Individuals currently undergoing treatment for pulmonary embolism or deep vein thrombosis
* Individuals with aortic (abdominal, thoracic) aneurysm
* Individuals with inflammatory bowel diseases
* Individuals currently undergoing hemodialysis
* Women with a past or family history of breast cancer.*1
* Women on estrogen replacement therapy
* Individuals unable to lay supine for 30-60 minutes
* Individuals with weight ≥300 lbs
* Individuals who are planning to move out of the area in the next 2 years
* Individuals who participated in another clinical trial in the past 3 months

Exclusion criteria via screening visit

* Individuals with Quick Dementia Rating System (QDRS) score ≥ 6.0
* Individuals who are regularly taking isoflavone supplements or eat soy product ≥ 2 times a week (by specific questionnaire)
* Individuals who do not agree to maintain isoflavone supplements or soy product intake described above during the study period.
* Individuals who have allergy or intolerance to soy isoflavones.
* Blood pressure (BP) - systolic BP ≥ 180 mmHg or diastolic BP ≥ 110 mmHg
* Heart rate ≥110 or ≤40
* Hemoglobin <10 g/dL
* HbA1c ≥ 7.5%
* Blood creatinine > 2.0 mg/dL
* Liver function tests > 2 X upper limit of normal
* Abnormal thyroid function (Thyroid Stimulating Hormone)
* Vitamin B12 levels ≤ 210 pg/mL
* Hematocrit <30%
* White blood cell count <3,000 or >15,000
* Platelet count <100,000 or >600,000
* Urinary protein ≥ + by dipstick
* Any condition or therapy which, in the opinion of the investigator, might pose a risk to the participant or make participation in the study not in the participant's best interest

In addition, individuals with the following condition will be excluded because these conditions do not allow subjects to undergo examinations the investigators proposed in the project:

* Those who are contraindicated for 3 Tesla (3T) structural brain magnetic resonance imaging (MRI) such as pacemakers.
* Atrial fibrillation because pulse wave velocity is not accurately measured.
* Hearing impairment which interferes with cognitive testing
* Vision impairment which interferes with cognitive testing

Exclusion criteria at structural brain MRI Any other conditions which, in the opinion of the investigator, might pose a risk to the participant or make participation in the study not in the participant's best interest

*1 Few studies have investigated the association of equol, a metabolite of soy isoflavone daidzein, with breast cancer. These studies reported no significant association of serum or urine equol with the risk of breast cancer. Dietary intake of soy and soy isoflavones is generally considered to have benefits for menopausal symptoms, cardiovascular health, bone health, and cancers of the breast and prostate. Observational studies show that soy consumption is associated with a reduced risk of many cancers including breast cancer. Moreover, a prospective cohort study of 6,000+ North American women with breast cancer showed that dietary intake of soy and isoflavones was associated with reduced all-cause mortality. However, there is little evidence to support that the use of supplements containing soy isoflavones or soy protein powder to reduce cancer risk. A recent large prospective cohort study in France reported that supplementation of soy isoflavones increased the risk of estrogen receptor-negative breast cancer, especially among women who had a history of breast cancer in first-degree relatives.

Exclusion criteria at the baseline visit

The investigators recruit subjects without dementia. Thus, at the initial screening by phone, the investigators exclude individuals whose score for the Telephone Interview for Cognitive Status is 22 and below. Then, at the screening visit, investigators will exclude individuals with a Quick Dementia Rating System score ≥ 6.0.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 369 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in arterial stiffness | Change from baseline in arterial stiffness at 12 months
  Arterial stiffness describes the rigidity of the arterial wall and is a significant predictor of cognitive decline. Arterial stiffness will be measured by pulse wave velocity (m/s) with a SphygmoCor device (Sydney, Australia). The range of pulse wave velocity is from 5 to 20 m/s.
Change in arterial stiffness | Change from baseline in arterial stiffness at 24 months
  Arterial stiffness describes the rigidity of the arterial wall and is a significant predictor of cognitive decline. Arterial stiffness will be measured by pulse wave velocity (m/s) with a SphygmoCor device (Sydney, Australia). The range of pulse wave velocity is from 5 to 20 m/s.

SECONDARY OUTCOMES:
Change in white matter lesion (WML) volume percent | Change from baseline in WML volume percent at 24 months
  WMLs are a significant predictor of cognitive decline. WMLs will be measured using an automated brain magnetic resonance imaging method. WML volume percent will be calculated by dividing WML volume by total brain volume as a percentage. The range of WML volume percent is from 0 to 4.2%.
Change in cognitive score measured by the Preclinical Alzheimer's Cognitive Composite-5 (PACC-5) score | Change from baseline in cognitive score measured by the PACC-5 at 12 months
  The PACC-5 is a composite neuropsychological measure optimized to detect subtle changes over time in cognitively unimpaired older adults. The range of PACC-5 score is from -3 to 3.
Change in cognitive score measured by the Preclinical Alzheimer's Cognitive Composite-5 (PACC-5) score. | Change from baseline in cognitive score measured by the PACC-5 at 24 months
  The PACC-5 is a composite neuropsychological measure optimized to detect subtle changes over time in cognitively unimpaired older adults. The range of PACC-5 score is from -3 to 3 where 3 represents better cognition.

OTHER OUTCOMES:
Change in NIH Toolbox (NIH-TB) cognition battery score | Change from baseline in NIH-TB cognition battery score at 12 months
  NIH-TB Cognition battery, comprised of computerized tests of fluid and crystallized cognitive abilities, via proctored iPad administration.
Change in NIH Toolbox (NIH-TB) cognition battery score | Change from baseline in NIH-TB cognition battery score at 24 months
  NIH-TB Cognition battery, comprised of computerized tests of fluid and crystallized cognitive abilities, via proctored iPad administration.
Changes in select brain markers other than white matter lesion (WML) volume percent | Change from baseline in brain markers other than WML volume percent at 24 months
  Brain markers other than WML volume percent will be measured using MRI, including cerebral blood flow, venous oxygenation, white matter organization lacunar infarct and cortical thickness.
Change in ultrasound measurements of carotid artery | Change from baseline in ultrasound measurements of carotid artery at 24 months
  Ultrasound measurements of carotid artery include carotid plaque and intima-media thickness. Investigators will use a high-resolution ultrasound system equipped with a variable frequency transducer (NextGen LOGIQ*e R7).
Change in select plasma biomarkers | Change from baseline in select plasma biomarkers at 24 months
  Plasma biomarkers of inflammation and endothelial function (C-reactive protein, intracellular adhesion molecule, vascular cell adhesion molecule, glial fibrillary acidic protein, neurofilament light) as well as amyloid-β40, amyloid-β42 and phosphorylated tau 181 will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Akira Sekikawa, MD, PhD, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Center for Clinical Trial & Data Coordination (CCDC), University of Pittsburgh, has rich experience as the Data Core (DC) for other NIH-funded studies, in reporting to and providing final datasets for an NIH Central Data Repository. The final dataset(s) will include demographic and clinical data at baseline, study arm assignment, and all primary and secondary outcomes for the ACE trial. The final dataset(s) will be completely de-identified. These data will be released to an NIH Central Data Repository no later than 1 year after the end of the clinical activity (final patient follow-up, etc.) or immediately after the main paper of the trial has been published, whichever comes first. The files available will include original copies of the case report forms, a detailed codebook of variable names, value labels, formats, missing data reports, and linkage files for samples. The analytic dataset may also include derived variables that were created during the analytic process.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The final dataset(s) will be completely de-identified. These data will be released to an NIH Central Data Repository no later than 1 year after the end of the clinical activity (final patient follow-up, etc.) or immediately after the main paper of the trial has been published, whichever comes first.
Access Criteria: Data Requestors must agree to the terms of the ACE Data Use Agreement (DUA) and will be asked to complete an online application for access to anonymized datasets. The agreement will be reviewed by the ACE Trial Steering Committee (SC).
  The ACE SC approval of the Data Requestor's Data Sharing Agreement request will trigger a process that allows access to the files described above and provides the requestor with an email notification of the review decision. All data and supporting documents selected by the project leadership for sharing will be made available for approved applicants to download. The review committee may require requestors to provide an annual update on their use of project data, to submit manuscripts for SC review and/or may revoke access for investigators who do not respond to annual update requests.

REFERENCES:
- [Background] Sekikawa A, Wharton W, Butts B, Veliky CV, Garfein J, Li J, Goon S, Fort A, Li M, Hughes TM. Potential Protective Mechanisms of S-equol, a Metabolite of Soy Isoflavone by the Gut Microbiome, on Cognitive Decline and Dementia. Int J Mol Sci. 2022 Oct 7;23(19):11921. doi: 10.3390/ijms231911921. PMID 36233223
- [Result] Sekikawa A, Wharton W, Murray-Krezan C, Wu M, Chang Y, Snitz BE, Coccari M, Yang S, Love ML, Cusick D, Wang R, Li M, Park C, Li J, DeConne TM, Smith C, Verble DD, Lancet MQ, Foroud T, Kim T, Nadkarni NK, Mettenburg JM, Zamora E, Lopez OL, Hughes TM. ACE trial design: Equol targeting estrogen receptor-beta in vascular and cognitive aging. Alzheimers Dement (N Y). 2025 Aug 18;11(3):e70144. doi: 10.1002/trc2.70144. eCollection 2025 Jul-Sep. PMID 40838083

DOCUMENTS (1):
  • Informed Consent Form (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT05741060/ICF_000.pdf